CLINICAL TRIAL: NCT00219544
Title: A Randomized, Placebo-Controlled Trial of the Efficacy and Safety of Pregabalin in the Treatment of Subjects With Peripheral Neuropathic Pain
Brief Title: Efficacy Study Measuring the Impact of Pregabalin on Peripheral Neuropathic Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081084
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-11

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Pregabalin (Lyrica)
- 2 (Experimental)
  Interventions: Drug: Pregabalin (Lyrica)
- 3 (Experimental)
  Interventions: Drug: Pregabalin (Lyrica)
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin (Lyrica) — pregabalin 150mg/day (75mg BID)
  Arms: 1
Drug: Pregabalin (Lyrica) — pregabalin 300 mg/day (150mg BID)
  Arms: 2
Drug: Pregabalin (Lyrica) — pregabalin 600/day (300mg BID)
  Arms: 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
This study will measure the impact of treatment with pregabalin in adult men and women who have a diagnosis of peripheral neuropathic pain (pain caused by a primary lesion of the peripheral nervous system such as Diabetic peripheral Neuropathy and Postherpetic Neuralgia).

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting a diagnosis of peripheral neuropathic pain, defined as pain caused by a lesion of the peripheral nervous system manifesting with sensory symptoms and signs, for at least 6 months at screening.
* At baseline, subjects must have completed at least 4 daily pain diaries and must have a mean weekly pain score equal or greater than 4.

Exclusion Criteria:

* Presence of any of the following diagnoses: Cervical or lumbo-sacral radiculopathy; Operated or non-operated chronic low back pain Carpal tunnel syndrome or any other entrapment-related neuropathic pain (defined as pain associated with focal nerve lesion produced by constriction or mechanical distortion of the nerve, within a fibrous or fibro-osseous tunnel, or by a fibrous band) ; Complex regional pain syndrome (type 1 and 2); Fibromyalgia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Canada (21):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Port Hope, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Granby, Quebec
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Lévis, Quebec
  - Pfizer Investigational Site, Mirabel, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Sherbrook, Quebec
  - Pfizer Investigational Site, Ste-Foy, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in Canada.
Pre-assignment Details: 405 subjects enrolled - 234 completed the single-blind phase. Subjects who responded (≥30% decrease in weekly mean pain score) during single-blind entered double-blind. 158 subjects assigned to study drug in double-blind phase. One subject in placebo group was randomized in error, not treated, not included as discontinuation;157 received treatment.
Groups:
- Pregabalin: subjects entered single-blind phase with 28 days of single-blind flexible pregabalin doses (150 to 600 mg/day), starting at 150 mg/day for ≥4 days, then dose adjustment as needed. Subjects who responded during the single-blind phase and were randomized to pregabalin entered the double-blind phase with 35 days of dose achieved at the end of the single-blind treatment phase.
- Placebo: subjects entered single-blind phase with 28 days of single-blind flexible pregabalin doses (150 to 600 mg/day), starting at 150 mg/day for ≥4 days, then dose adjustment as needed. Subjects who responded during the single-blind phase and were randomized to placebo received pregabalin 150 mg for 7 days and then placebo for 28 days.
Period: Single Blind Treatment Period
Arm/Group | Pregabalin | Placebo
Started | 256 | 0
Completed | 234 | 0
Not Completed | 22 | 0
Not completed — Lack of Efficacy | 5 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Investigator decision to withdraw | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Double Blind Treatment Period
Arm/Group | Pregabalin | Placebo
Started | 80 | 77
Completed | 80 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 128

OUTCOME MEASURES:

1. Primary Outcome: Neuropathic Pain in Subjects With Peripheral Neuropathic Pain Conditions During the Double-blind Phase
Description: Pain score end of Double-Blind treatment = mean of last 7 available pain scores from daily pain diary while on Double-Blind treatment. A Daily Pain Rating Score : 11- point numerical scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: 9 weeks
Population: Full Analysis Set (FAS) = Intent-to-Treat (ITT) population, defined as all subjects who are randomized into the Double-Blind treatment phase, who receive at least one dose of Double-Blind study medication and complete at least one postrandomization efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale | 2.84 (0.18) | 3.62 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; The study is powered to detect clinically significant difference of 1.2 between treatment groups in mean pain score at end of treatment. The statistical sample size calculation requires a total of 144 subjects to complete the Double-Blind phase of the study: a sample size of 72 in each treatment group will have 90% power to detect a difference in treatment mean pain scores of 1.2 assuming that the common standard deviation is 2.2 using a two group t-test with a 0.05 two-sided significance level; Test type: Superiority or Other; p = 0.0018, ANCOVA; Mean Difference (Net) = -0.78, 95% CI [-1.27 to -0.30], Standard Error of Mean 0.25 — Difference = pregabalin minus placebo

2. Secondary Outcome: Weekly Mean Pain Scores During the Single-blind Treatment Phase
Description: Pain score at Week 0 and Week 4, end of single-bind treatment. Mean of last 7 available pain scores from daily pain diary while on single-blind treatment. A Daily Pain Rating Score : 11- point numerical scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: 0 and 4 weeks
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Pregabalin: subjects entered single-blind phase with 28 days of single-blind flexible pregabalin doses (150 to 600 mg/day) for ≥4 days, then dose adjustment as needed.
Arm/Group | Pregabalin
Number analyzed (Participants) | 255
score on scale
  Week 0 - Baseline | 6.29 (1.43)
  Week 4 - end of single-blind treatment | 3.79 (2.11)

3. Secondary Outcome: Weekly Mean Pain Scores During the Double Blind Treatment Phase
Description: Mean Pain scores for weeks 4, 5, 6, 7, 8 and 9. Mean of last 7 available pain scores from daily pain diary while on single-blind treatment. A Daily Pain Rating Score : 11-point numerical scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: Week 4 - 9
Population: FAS population.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale
  Week 4 (n=73, 70) | 2.68 (1.29) | 2.49 (1.23)
  Week 5 (n=70,64) | 2.62 (1.48) | 3.14 (1.41)
  Week 6 (n=66,63) | 2.75 (1.76) | 3.40 (1.49)
  Week 7 (n=60,56) | 2.53 (1.80) | 3.20 (1.45)
  Week 8 (n=63,53) | 2.51 (1.59) | 3.16 (1.54)
  Week 9 (n=67,58) | 2.80 (1.80) | 3.29 (1.52)

4. Secondary Outcome: Change in Pain Scores During Double Blind Treatment Phase
Description: Change in Mean Pain score = Mean of last 7 available pain scores from daily pain diary while on single-blind treatment. A Daily Pain Rating Score : 11-point numerical scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: 9 weeks
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale
  Change from randomization to Week 5 (n=70, 64) | -0.01 (0.15) | 0.71 (0.16)
  Change from randomization to Week 6 (n=66, 63) | 0.08 (0.16) | 1.05 (0.16)
  Change from randomization to Week 7 (n=60, 56) | -0.06 (0.16) | 0.87 (0.17)
  Change from randomization to Week 8 (n=63,53) | -0.10 (0.16) | 0.83 (0.17)
  Change from randomization to Week 9 (n=67,58) | 0.14 (0.15) | 0.84 (0.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0010, ANCOVA; Mean Difference (Net) = -0.72, 95% CI [-1.15 to -0.30], Standard Error of Mean 0.22 — pregabalin minus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = -0.97, 95% CI [-1.41 to -0.53], Standard Error of Mean 0.22 — pregabalin minus placebo
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 7; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = -0.93, 95% CI [-1.39 to -0.47], Standard Error of Mean 0.23 — pregabalin minus placebo
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = -0.93, 95% CI [-1.39 to -0.47], Standard Error of Mean 0.23 — pregabalin minus placebo
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 9; Test type: Superiority or Other; p = 0.0022, ANCOVA; Mean Difference (Net) = -0.69, 95% CI [-1.14 to -0.25], Standard Error of Mean 0.23 — pregabalin minus placebo

5. Secondary Outcome: Number of Subjects With >= 30% Reduction in Mean Pain Score During Single-blind Treatment
Description: Responders = ≥30% reduction in mean pain score at end of single-blind treatment phase compared to weekly mean pain score at baseline. Mean of last 7 available pain scores from daily pain diary while on single-blind treatment. A Daily Pain Rating Score : 11-point numerical scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: Week 4 (end of single-blind treatment phase)
Population: 256 subjects entered the single-blind treatment phase, one subject did not have enough DPRS assessments for calculation.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 255
participants
  Responders | 165
  Non-Responders | 90

6. Secondary Outcome: Mean Pain Score for Responders at End of Single-blind Treatment Phase. Change From Baseline of Mean of Last 7 Available Pain Scores From Daily Pain Diary While on Single-blind Treatment.
Description: Daily Pain Rating Score:11-point numerical scale 0 ("no pain") to 10 ("worst possible pain"). Responders = ≥30% reduction in mean pain score at end of single-blind treatment phase compared to weekly mean pain score at baseline.
Time Frame: Week 4
Population: number of subjects that can be analyzed for Change from Baseline at End of Single Blind.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 165
score on scale | -3.60 (1.32)

7. Secondary Outcome: Mean Pain Score for Non-responders at End of Single-blind Treatment Phase
Description: Change from baseline of mean of last 7 available pain scores from daily pain diary while on single-blind treatment. Daily Pain Rating Score:11-point numerical scale 0 ("no pain") to 10 ("worst possible pain"). Non-Responders = <30% reduction in mean pain score at end of single-blind treatment phase compared to weekly mean pain score at baseline.
Time Frame: Week 4
Population: number of subjects that can be analyzed for Change from Baseline at End of Single Blind.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 90
score on scale | -0.49 (0.95)

8. Secondary Outcome: Categorized Daily Pain Score
Description: Mean number of days in each pain category. DPRS Daily Pain Rating Score Categories: No pain (score 0), Mild pain (scores 1-3), Moderate pain (scores 4-6), Severe pain (scores 7-10)
Time Frame: Week 9
Population: Number of subjects analyzed for each pain category.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 73 | 71
days
  No pain | 3.3 (7.6) | 0.9 (3.1)
  Mild pain | 19.5 (12.1) | 17.4 (11.9)
  Moderate pain | 7.4 (9.5) | 8.6 (8.3)
  Severe pain | 1.2 (2.8) | 1.7 (4.5)

9. Secondary Outcome: Time to Meaningful Increase in Pain During Double-blind Treatment Phase (Number of Participants)
Description: Number of participants who experienced a meaningful increase in pain also includes participants who took rescue medication for pain due to peripheral neuropathic pain or discontinued from the study .
Time Frame: Week 9
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 80 | 77
participants | 28 | 28

10. Secondary Outcome: Mean Sleep Interference Score
Description: Mean Sleep Interference (SI) score at end of Double-Blind treatment = mean of last 7 available SI scores from daily SI diary while on Double-Blind treatment. Daily SI rating scale (DSIS) consists of an 11-point numerical scale : Zero means "pain does not interfere with sleep" and 10 means "pain completely interferes with sleep."
Time Frame: Week 9
Population: FAS population.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale | 1.81 (0.17) | 2.52 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0031, ANCOVA; Median Difference (Net) = -0.71, 95% CI [-1.18 to -0.24], Standard Error of Mean 0.24

11. Secondary Outcome: Weekly Mean Sleep Interference Scores During the Single-Blind Treatment Phase
Description: Sleep Interference (SI) score at Week 0 and Week 4, end of single-bind treatment. Mean of last 7 available SI scores from daily SI diary while on single-blind treatment. Daily SI rating scale (DSIS) consists of an 11-point numerical scale : Zero means "pain does not interfere with sleep" and 10 means "pain completely interferes with sleep."
Time Frame: 0 and 4 weeks
Population: Last observation carried forward (LOCF) approach for patients who do not complete the study will be adopted. This is defined as the mean of the last 7 diary scores while on Double-Blind study drug, up to and including the day after the last day on drug (excluding the taper phase).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 255
score on scale
  Week 0 - Baseline | 4.80 (2.44)
  Week 4 - end of single-blind treatment | 2.72 (2.42)

12. Secondary Outcome: Weekly Mean Sleep Interference Scores During the Double Blind Treatment Phase
Description: Mean Sleep Interference scores for weeks 4, 5, 6, 7, 8 and 9. Mean of last 7 available SI scores from daily SI diary while on single-blind treatment. Daily SI rating scale (DSIS) consists of an 11-point numerical scale : Zero means "pain does not interfere with sleep" and 10 means "pain completely interferes with sleep."
Time Frame: Week 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale
  Week 4 (n=73, 70) | 1.68 (1.57) | 1.62 (1.61)
  Week 5 (n=70,64) | 1.76 (1.61) | 2.24 (1.79)
  Week 6 (n=66,63) | 1.85 (1.81) | 2.53 (1.69)
  Week 7 (n=60,56) | 1.66 (1.63) | 2.38 (1.75)
  Week 8 (n=63,53) | 1.59 (1.57) | 2.36 (1.79)
  Week 9 (n=67,58) | 1.66 (1.74) | 2.40 (1.86)

13. Secondary Outcome: Change in Sleep Interference Scores During Double Blind Treatment Phase
Description: Change in Mean SI score: Mean SI score at observation minus mean SI score at week 4. Mean SI Score = mean of last 7 available SI scores from daily SI diary while on single-blind treatment. Daily SI rating scale (DSIS) is 11-point numerical scale : Zero means "pain does not interfere with sleep" and 10 means "pain completely interferes with sleep."
Time Frame: 9 weeks
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 73 | 70
score on scale
  Change from randomization to Week 5 (n=70, 64) | 0.07 (0.15) | 0.59 (0.16)
  Change from randomization to Week 6 (n=66, 63) | 0.10 (0.16) | 0.97 (0.16)
  Change from randomization to Week 7 (n=60, 56) | -0.03 (0.16) | 0.78 (0.17)
  Change from randomization to Week 8 (n=63,53) | -0.13 (0.16) | 0.72 (0.17)
  Change from randomization to Week 9 (n=67,58) | -0.01 (0.15) | 0.73 (0.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0177, ANCOVA; Mean Difference (Net) = -0.52, 95% CI [-0.94 to -0.09], Standard Error of Mean 0.22 — pregabalin minus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = -0.87, 95% CI [-1.31 to -0.44], Standard Error of Mean 0.22 — pregabalin minus placebo
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 7; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Net) = -0.82, 95% CI [-1.28 to -0.36], Standard Error of Mean 0.23 — pregabalin minus placebo
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Net) = -0.85, 95% CI [-1.31 to -0.39], Standard Error of Mean 0.23 — pregabalin minus placebo
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 9; Test type: Superiority or Other; p = 0.0011, ANCOVA; Mean Difference (Net) = -0.74, 95% CI [-1.18 to -0.30], Standard Error of Mean 0.22 — pregabalin minus placebo

14. Secondary Outcome: Intensity of Neuropathic Pain -Visual Analog Scale (NeP - VAS)
Description: Change in Scale from randomization to Week 9. Scale to measure Neuropathic Pain -Visual Analog Scale (NeP - VAS): the subject places a mark on the VAS scale (0 to 100) where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Week 4, Week 9
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 73
scores on a scale | 6.9 (2.4) | 15.9 (2.5)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0069, ANCOVA; Mean Difference (Net) = -9.0, 95% CI [-15.5 to -2.5], Standard Error of Mean 3.3

15. Secondary Outcome: Change in Hospital Anxiety and Depression Scale Responses
Description: Mean Change from Randomization in Score from Hospital Anxiety and Depression Scale (HADS): 2 subscales, measuring anxiety (HADS-A)and depression (HADS-D). 7 items in each subscale assessed on a scale of 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). which yields the score ranging 0-21.
Time Frame: Week 9
Population: FAS population
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale
  HADS-A | -0.1 (0.3) | 1.2 (0.3)
  HADS-D | -0.4 (0.3) | 0.8 (0.3)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; HADS-A; Test type: Superiority or Other; p = 0.0023, ANCOVA; Mean Difference (Net) = -1.3, 95% CI [-2.1 to -0.5], Standard Error of Mean 0.4 — pregabalin minus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; HADS-D; Test type: Superiority or Other; p = 0.0013, ANCOVA; Mean Difference (Net) = -1.2, 95% CI [-1.9 to -0.5], Standard Error of Mean 0.4 — pregabalin minus placebo

16. Secondary Outcome: Change in Pain Treatment Satisfaction Scale (PTSS)
Description: Mean Change: score from observation minus score from randomization: PTSS "Impact" module of 8-items & "Satisfaction" module of 6-items; item scores 1-5.
  Mean score for each module transformed onto scale 0- 100, where score 0 =worst possible response and score 100
  =best possible response: Score =[(5 - mean non-missing items)*100]/4.
Time Frame: Week 9
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 73 | 70
score on scale
  impact of current pain medication | -1.96 (2.53) | -7.95 (2.60)
  satisfaction with current pain medication | -1.86 (2.04) | -8.35 (2.09)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Impact; Test type: Superiority or Other; p = 0.0828, ANCOVA; Mean Difference (Net) = 5.98, 95% CI [-0.79 to 12.75], Standard Error of Mean 3.42 — pregabalin minus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Satisfaction; Test type: Superiority or Other; p = 0.0197, ANCOVA; Mean Difference (Net) = 6.49, 95% CI [1.05 to 11.94], Standard Error of Mean 2.75 — pregabalin minus placebo

17. Secondary Outcome: Patient Global Impression of Change (PGIC) Categories by Number of Subjects
Description: Number of subjects that responded to PGIC Categories. PGIC is a subject-rated instrument that measures change in the subject's overall status on a 7-point scale. Scores range from
  1 (very much improved) to 7 (very much worse).
Time Frame: Week 9
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
participants
  Very much improved | 21 | 12
  Much improved | 35 | 32
  Minimally improved | 15 | 17
  No change | 6 | 7
  Minimally worse | 0 | 6
  Much worse | 1 | 0
  Very much worse | 0 | 1
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; The distribution of the responses to the PGIC at EOT was compared between the 2 treatment groups using the 7 categories of the PGIC; Test type: Superiority or Other; p = 0.0278, Mantel Haenszel

18. Secondary Outcome: Change in Modified Brief Pain Inventory (mBPI) for Pain Interference or Pain Severity.
Description: Mean Change from Randomization: score at mBPI observation minus score at randomization. mBPI is extent to which pain interferes with daily activities on a 0 (no interference) to 10 (completely interfered) scale.
Time Frame: Week 9
Population: FAS population
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale
  Pain interference | 0.16 (0.19) | 0.92 (0.20)
  Pain severity | 0.29 (0.19) | 1.06 (0.19)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Pain interference; Test type: Superiority or Other; p = 0.0049, ANCOVA; Mean Difference (Net) = -0.76, 95% CI [-1.28 to -0.23], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Pain severity; Test type: Superiority or Other; p = 0.0037, ANCOVA; Mean Difference (Net) = -0.77, 95% CI [-1.29 to -0.25], Standard Error of Mean 0.26

19. Secondary Outcome: Change in Euro Quality of Life (EQ-5D) Health State Profile and Visual Analog Scale Components
Description: two components to the EQ-5D: a Health State Profile (scores from five domains are used to calculate the utility score :0 refers to dead and a score of 1 refers to perfect health) and a Visual Analogue Scale (VAS) (0 represents the worst imaginable health state and 100 represents the best imaginable health state)
Time Frame: Week 9
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 75
score on scale
  Health State Profile | -0.01 (0.02) | -0.07 (0.02)
  Visual Analog Scale | -0.03 (1.83) | -2.09 (1.89)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Health State Profile; Test type: Superiority or Other; p = 0.0719, ANCOVA; Mean Difference (Net) = 0.05, 95% CI [-0.00 to 0.11], Standard Error of Mean 0.03 — pregabalin minus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Visual Analog Scale; Test type: Superiority or Other; p = 0.4180, ANCOVA; Mean Difference (Net) = 2.07, 95% CI [-2.96 to 7.10], Standard Error of Mean 2.54 — pregabalin minus placebo

ADVERSE EVENTS:
Groups:
- Pregabalin Single-blind Phase: subjects entered single-blind phase with 28 days of single-blind flexible pregabalin doses (150 to 600 mg/day) for ≥4 days, then dose adjustment as needed.
- Pregabalin Double-blind Phase: subjects entered single-blind phase with 28 days of single-blind flexible pregabalin doses (150 to 600 mg/day) for ≥4 days, then dose adjustment as needed. Subjects who responded during the single-blind phase and were randomized to pregabalin entered the double-blind phase with 35 days of dose achieved at the end of the single-blind treatent phase.
- Placebo Double-blind Phase: subjects entered single-blind phase with 28 days of single-blind flexible pregabalin doses (150 to 600 mg/day) for ≥4 days, then dose adjustment as needed. Subjects who responded during the single-blind phase and were randomized to placebo received pregabalin 150 mg for 7 days and then placebo for 28 days.
Arm/Group | Pregabalin Single-blind Phase | Pregabalin Double-blind Phase | Placebo Double-blind Phase
Serious Adverse Events (participants affected / at risk) | 1 | 0 | 0
Other Adverse Events (participants affected / at risk) | 196 | 33 | 29
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pregabalin Single-blind Phase | Pregabalin Double-blind Phase | Placebo Double-blind Phase
Pneumonia (Infections and infestations) | 1/256 (1) | 0/80 (0) | 0/77 (0)
Sepsis (Infections and infestations) | 1/256 (1) | 0/80 (0) | 0/77 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/256 (1) | 0/80 (0) | 0/77 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pregabalin Single-blind Phase | Pregabalin Double-blind Phase | Placebo Double-blind Phase
Asthenia (Surgical and medical procedures) | 24/256 | 5/80 | 2/77
Headache (General disorders) | 24/256 | 5/80 | 6/77
Pain (General disorders) | 7/256 | 3/80 | 5/77
Constipation (Gastrointestinal disorders) | 13/256 | 1/80 | 0/77
Dry mouth (Gastrointestinal disorders) | 46/256 | 0/80 | 0/77
Nausea (Gastrointestinal disorders) | 19/256 | 4/80 | 3/77
Peripheral edema (Metabolism and nutrition disorders) | 35/256 | 6/80 | 2/77
Arthralgia (Musculoskeletal and connective tissue disorders) | 8/256 | 2/80 | 5/77
Weight gain (Metabolism and nutrition disorders) | 16/256 | 5/80 | 1/77
Balance Disorder (Nervous system disorders) | 18/256 | 2/80 | 1/77
Dizziness (Nervous system disorders) | 90/256 | 7/80 | 8/77
Euphoria (Nervous system disorders) | 13/256 | 1/80 | 0/77
Somnolence (Nervous system disorders) | 48/256 | 3/80 | 2/77
Thinking abnormal (Nervous system disorders) | 29/256 | 1/80 | 0/77
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 17/256 | 7/80 | 8/77
Abnormal vision (Eye disorders) | 23/256 | 2/80 | 1/77
Diarrhea (Gastrointestinal disorders) | 12/256 | 4/80 | 2/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.